CLINICAL TRIAL: NCT03231254
Title: Differences in Predicted Therapeutic Outcome of Oral Appliance and Optimal Protrusion Position Determined by Remotely Controlled Mandibular Positioner (RCMP) With Overnight PSG in Quebec Versus Shenyang Patients With OSA
Brief Title: Differences in Predicted Therapeutic Outcome of Oral Appliance Determined by RCMP in Quebec Versus Shenyang Patients With OSA.
Acronym: RCMP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Hospital of China Medical University (Other)
Collaborators: Laval University (Other)
Responsible Party: Principal Investigator, Wenyang Li, Medical doctor, First Hospital of China Medical University
Other Study IDs: AF-SOP-07-1.0-01
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Remotely Controlled Mandibular Positioner

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Chinese patients with OSA
  Interventions: Device: Remotely Controlled Mandibular Positioner (RCMP)
- Canada patients with OSA
  Interventions: Device: Remotely Controlled Mandibular Positioner (RCMP)

INTERVENTIONS:
Device: Remotely Controlled Mandibular Positioner (RCMP) — RCMP device can accurately identify patients who are likely to be successful OA candidates. With a temporary dental appliance connected to a RCMP, the mandible could be progressively, mildly and precisely protruded in only anterior-posterior dimension, under the monitor of PSG, without disturbing sleep, until obstructive apneas and hypopneas were eliminated, particularly in REM sleep while supine. Besides, RCMP device can also determine the optimal therapeutic level of mandibular protrusion during sleep.

SUMMARY:
Study Objective: To explore the differences in predicted therapeutic outcome of OA and optimal protrusion position determined by Remotely Controlled Mandibular Positioner (RCMP) with overnight PSG in Quebec versus Shenyang patients with OSA.

Design: A prospective, inter-ethnic pilot study. Setting: Two Standard sleep disorder clinical care in Quebec (Canada) and Shenyang (China), with oral appliance titration tests performed in sleep laboratory.

Participants: Consecutive specific OSA patients, who are potential candidates for treatment of OSA with an oral appliance (n=100, 50 Canadian, 50 Chinese), will be recruited from a sleep center or respirologists, psychiatrists, otolaryngologist and dentists practicing with broad inclusion criteria (age: 20-75 years, AHI:15-50/h; BMI<40 kg/m2).

Interventions: A mandibular protrusive titration study in the PSG lab using a RCMP not only predicts the eventual therapeutic outcome but also prospectively determines Optimal Protrusive Position (OPP) for participants predicted to be therapeutically successful with OA therapy. One goal of this study is to identify OA favorable candidates by physicians using prospectively and explicitly designed criteria. Analyses of the predicted therapeutic outcome of OA and OPP between the two ethnic populations (patients in Quebec and Shenyang) will be processed after matching for OSA severity.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of OSAS (AHI>15/h) announced by a sleep recording; mean oxygen saturation >90%; mandibular range of motion >5 mm; adequate dentition: ≥10 upper and 10 lower teeth.

Exclusion Criteria:

* (1). Body mass index 40 kg/m2 or greater; (2).Inability to tolerate overnight polysomnography in sleep lab; (3).>50% of observed sleep apneas being central; (4). Other sleep disorders such as insomnia, narcolepsy, chronic sleep deficiency, periodic limb movement disorder or restless legs syndrome; (5). Those with severe pharyngeal obstruction on physical exam (pharyngeal grade more than II); (6).severe nasal obstruction.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Research participants will be respectively recruited from Sleep Centre of IOCPQ of Laval (Quebec, Canada) and CMU first affiliated hospital (Shenyang, China), which receives the majority of referrals from respirologists, psychiatrists, otolaryngologists and dentists practicing in Quebec and Shenyang City. Consecutive patients between 20 and 75 years of age, satisfying the pre-mentioned inclusion will be considered eligible to our study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-10-20 (Estimated); Study Completion 2017-10-29 (Estimated)

PRIMARY OUTCOMES:
The differences of predicted therapeutic outcome of OA between two groups. | 2017.7-2017.11
  To identify and compare the number of OA favorable candidates by physicians using prospectively and explicitly designed criteria in both groups.

SECONDARY OUTCOMES:
The differences of optimal protrusion position determined by Remotely Controlled Mandibular Positioner (RCMP) with overnight PSG in Quebec versus Shenyang patients with OSA. | 2017.7-2017.11

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, PhD, Principal Investigator — First Hospital of China Medical University; Frederic Series, master, Study Director — Pneumologue Institut Universitaire de Cardiologie et de Pneumologie de Québec
Locations (2):
- Frederic Series, Québec, Quebec, Canada
- Wenyang Li, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Remmers J, Charkhandeh S, Grosse J, Topor Z, Brant R, Santosham P, Bruehlmann S. Remotely controlled mandibular protrusion during sleep predicts therapeutic success with oral appliances in patients with obstructive sleep apnea. Sleep. 2013 Oct 1;36(10):1517-25, 1525A. doi: 10.5665/sleep.3048. PMID 24082311
- [Derived] Li WY, Masse JF, Gakwaya S, Zhao Z, Wang W, Series F. Differences in Predicted Therapeutic Outcome of Mandibular Advancement Determined by Remotely Controlled Mandibular Positioner in Canadian and Chinese Apneic Patients. Nat Sci Sleep. 2022 Sep 8;14:1611-1622. doi: 10.2147/NSS.S377758. eCollection 2022. PMID 36105925